CLINICAL TRIAL: NCT00510991
Title: Non Invasive Ventilation in Acute Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
Keywords: ASTHMA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): NIPPV
  Interventions: Device: nippv

INTERVENTIONS:
Device: nippv

SUMMARY:
The aim of this study is to compare the efficacy of noninvasive positive pressure ventilation versus best medical therapy in patients with acute severe asthma

DETAILED DESCRIPTION:
In the past, the mainstay of treatment for patients progressing to respiratory failure from acute asthma was intubation and mechanical ventilation. Newer strategies to prevent these intubations to prevent the inherent complications are being explored in form of various pharmacological means like heliox, magnesium sulfate etc. Non pharmacological strategies among which non invasive positive pressure ventilation (NIPPV) is one of the most challenging after showing success in patients with chronic obstructive airway disease (COPD) and cardiogenic pulmonary edema.

Data on efficacy of NIPPV in the management of AA is sparse but has the potential to improve the management of acute severe asthma. Noninvasive ventilation merits further studies in patients with AA, and some consensus panels have suggested that its widespread application in patients with asthma await such trials.The role of NIPPV is not yet clear and needs further studies and keeping this in view we planned this study to study the role of NIPPV in the management of acute asthma.

ELIGIBILITY:
Inclusion Criteria:

1. History of asthma of at least 1 year
2. FEV1 < 50% of predicted (by age, height, and gender) or FEV1 < 200 L/minute
3. Respiratory rate > 30 breaths/min
4. All patients judged by the attending physician as having an acute attack of asthma ( Inability to speak in sentences in one breath, SaO2 < 92% ,pulsus paradoxus > 10 mm of Hg) -

Exclusion Criteria:

1. Smoking history of > 10 years
2. Chronic obstructive pulmonary disease
3. Endotracheal intubation
4. Room air saturation < 88 % or arterial PaO2 < 55 mm of Hg
5. Hemodynamic instability defined as systolic BP < 90 mm Hg
6. Altered state of consciousness
7. Congestive heart failure
8. Ischemic heart disease
9. Upper airway obstruction
10. Facial deformity
11. Pregnancy
12. Pulmonary infiltrates consistent with pulmonary edema or pneumonia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in lung function defined as an increase of at least 50% in FEV1 as compared to baseline value on admission or an increase in FEV1 to > 60% of predicted value | Time to discharge
Intensive care unit length of stay | Time to discharge
Hospital length of stay | Time to discharge

SECONDARY OUTCOMES:
Improvement in the clinical status | Time to discharge
Disappearance of pulsus paradoxus | Time to discharge
Improvement in arterial blood gases | Time to discharge
Improvement in oxygen saturation | Time to discharge
Requirements of FiO2 , medications. | Time to discharge
Need for mechanical ventilation | Time to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alok Nath, MD, Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Gupta D, Nath A, Agarwal R, Behera D. A prospective randomized controlled trial on the efficacy of noninvasive ventilation in severe acute asthma. Respir Care. 2010 May;55(5):536-43. PMID 20420722